CLINICAL TRIAL: NCT03424473
Title: Expanded Access Use of Tucatinib for HER2+ Metastatic Breast Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ONT-380-014
Record Dates: First submitted 2018-01-31; First posted 2018-02-07 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

Keywords: tucatinib; Breast Cancer; ARRY-380; ONT-380; HER2 Positive Breast Carcinoma; HER2 Positive Locally Advanced Breast Cancer; HER-2 Positive Breast Cancer; HER-2 Positive Locally Advanced Breast Cancer; Recurrent Breast Carcinoma; Stage IV Breast Cancer; Metastatic Breast Cancer; Breast Carcinoma; Metastatic Malignant Neoplasm in the Brain; Brain Metastases in Breast Cancer; Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases | interventions — tucatinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Tucatinib

SUMMARY:
Physicians interested in requesting a single patient IND should contact Seattle Genetics' Medical Information (medinfo@seagen.com).

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult